CLINICAL TRIAL: NCT03728153
Title: MAMBO: Measuring Ambulation, Motor, and Behavioral Outcomes With Post-Stroke Fluoxetine in Tanzania
Brief Title: Measuring Ambulation, Motor, and Behavioral Outcomes With Post-Stroke Fluoxetine in Tanzania
Acronym: MAMBO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Muhimbili University of Health and Allied Sciences (Other)
Responsible Party: Principal Investigator, Farrah Mateen, Associate Professor, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018P001693
Record Dates: First submitted 2018-10-29; First posted 2018-11-01 (Actual); Results first posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Acute Stroke; Stroke, Ischemic
Keywords: Motor recovery
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — Fluoxetine; Tablets

STUDY DESIGN:
Intervention Model Description: Phase II study of one dose
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- 20mg dose (Experimental): Fluoxetine 20 MG Oral Tablet
  Interventions: Drug: Fluoxetine 20 MG Oral Tablet

INTERVENTIONS:
Drug: Fluoxetine 20 MG Oral Tablet — Once-daily dosing for 90 days
  Other Names: Prozac 20 MG Oral Tablet

SUMMARY:
This is a phase II, randomized study of 120 adults age 18 or above who will prescribed 20mg daily Fluoxetine for 90 days following acute, ischemic stroke.

DETAILED DESCRIPTION:
This is a prospective, phase II study of fluoxetine for motor recovery post-stroke in adults with new-onset ischemic stroke in urban Tanzania. Participants will be enrolled at the Muhimbili National Hospital (MNH) in Dar Es Salaam after confirmation of exclusion and inclusion criteria, including a head CT. Participants will be enrolled within 21 days of acute, ischemic stroke. The study will utilize a novel method for monitoring patient medication adherence: electronic pill bottles that can record medication use events. The primary goals of this study are to assess the safety and tolerability of fluoxetine post-stroke to evaluate the feasibility of conducting a larger, phase III study in the future.

Vital status will be monitored throughout the study's enrollment period. At enrollment, participants will have cognitive tests administered, receive lumbar puncture, and receive an MRI brain. After discharge from the hospital, participants will be seen at 30-, 60-, and 90-days post-enrollment for an in-person study visit. At each time point, investigators will draw 10-15 mL of blood; download medication adherence data from participants' electronic pill bottles; and inquire about adverse events and evaluate patient disability through the modified Rankin Scale. If participants stop taking their daily pill, stroke specific reasons for non-adherence will be inquired including dysphagia, self-administration, and other concerns.

Primary assessments will be for safety and tolerability, as well as measurement of the Fugl-Meyer Motor Scale. Medication use data will also be collected through the electronic pill bottle, which will be returned to study investigators. As secondary assessments, the PHQ-9, and the Asberg Depressive Symptom Questionnaire will be administered. All 90-day assessments will be administered by senior site investigators, who will take a final 10-15mL blood draw to test for serum sodium and liver enzymes, possible adverse events related to long-term fluoxetine use, conduct a second MRI brain, evaluate participant mRS, and inquire about tolerability issues. Completion of the 90-day visit and associated assessments is considered the study endpoint.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is 18 years of age or older
2. Participant has experienced a CT-confirmed ischemic stroke w/in 21 days of enrollment

Exclusion Criteria:

1. NIH Stroke Scale Score >20 points
2. Unconscious at presentation
3. Hemorrhagic conversion of ischemic infarct
4. transient ischemic symptoms <24h,
5. Current antidepressant or psychoactive drug use (e.g. SSRI, monoxidase amine inhibitor, benzodiazepine).
6. Current pregnancy.
7. History of recent head trauma.
8. Baseline motor deficits from other etiologies including prior stroke.
9. Dysphagia preventing the swallowing of a pill.
10. Hyponatremia (<125 mmol/L), hepatic impairment as defined by a serum alanine aminotransferase (ALT) of >120 U/L.
11. Renal impairment as defined by a creatinine >180 micromol/L or GFR <30mL/min/1.73m2.
12. Patients who are moribund for other reasons and unlikely to survive to 90 days will also be excluded from participation.
13. Contraindication to MRI (e.g. piercings/tattoos, electronic/metallic implants, claustrophobia)
14. Contraindication to lumbar puncture (e.g. infection at site of needle insertion, evidence of elevated ICP, coagulopathy/thrombocytopenia or use of therapeutic anticoagulation, or a history of LP complications).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-11-26 (Actual); Primary Completion 2021-01-06 (Actual); Study Completion 2021-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Farrah J Mateen, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Muhimbili National Hospital, Dar es Salaam, Tanzania

IPD SHARING:
Plan to Share IPD: No
Contingent upon the requirements of the Tanzanian National Medical Institute for Research

REFERENCES:
- [Background] Vogel AC, Okeng'o K, Chiwanga F, Ismail SS, Buma D, Pothier L, Mateen FJ. MAMBO: Measuring ambulation, motor, and behavioral outcomes with post-stroke fluoxetine in Tanzania: Protocol of a phase II clinical trial. J Neurol Sci. 2020 Jan 15;408:116563. doi: 10.1016/j.jns.2019.116563. Epub 2019 Nov 6. PMID 31731111

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 20mg Dose
Started | 34
Completed | 32
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | 20mg Dose
Number analyzed (Participants) | 34
Age, Continuous [Mean (Full Range); unit: years] | 52 [21 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 34
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Tanzania | 34

OUTCOME MEASURES:

1. Primary Outcome: Serum Sodium Concentration
Description: Serum Sodium Concentration was measured in mmol/L. Hyponatremia was considered as <125 mmol/L.
Time Frame: 90 days following acute, ischemic stroke
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | 20mg Dose
Number analyzed (Participants) | 32
mmol/L | 138.7 (2.9)

2. Primary Outcome: Serum Alanine Aminotransferase (ALT)
Description: Hepatic impairment was measured by elevation of hepatic enzyme (serum alanine aminotransferase; ALT) of >120 U/L
Time Frame: 90 days
Measure: Mean (Full Range); unit: U/L
Arm/Group | 20mg Dose
Number analyzed (Participants) | 32
U/L | 28 [10 to 134]

3. Secondary Outcome: Fugl-Meyer Motor Scale Score for Assessment of Motor Function After Stroke
Description: The Fugl Meyer motor scale is used to assess post-stroke motor recovery in stroke patients. It is scored on a scale from 0 to 100, with lower scores indicating greater disability. It evaluates both lower and upper extremities for motor performance: 66 points are allocated to the upper extremities, 34 to the lower extremities. The two extremities are summed to achieve the total score.
Time Frame: 90 days following acute, ischemic stroke
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 20mg Dose
Number analyzed (Participants) | 32
score on a scale | 62.7 (28.1)

4. Secondary Outcome: Montgomery-Asberg Depression Rating Scale
Description: 10-item questionnaire used to evaluate the severity of a patient's depressive symptoms. Each item is scored on a scale from 0 to 6, the scores are summed, and the total score (0 to 60 points) is reported. The greater the score, the more severe the degree of depression.
Time Frame: 90 days following acute, ischemic stroke
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 20mg Dose
Number analyzed (Participants) | 32
units on a scale | 5.6 (5.5)

5. Secondary Outcome: Modified Rankin Scale
Description: Validated instrument for measuring the degree of disability in stroke patients. The modified Rankin Scale is based on a physicians subjective evaluation. The scale ranges from 0, indicating perfect health, to 6, indicating that the patient is dead.
Time Frame: 90 days following acute, ischemic stroke
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | 20mg Dose
Number analyzed (Participants) | 32
score on a scale | 2 [1 to 3]

6. Secondary Outcome: The Patient Health Questionnaire-9 (PHQ-9) Scale for Measuring Depression
Description: The PHQ-9 is a validated 9-point questionnaire for measuring depression symptom severity. Each question is scored from 0-3. Answers are summed and the total score (0 to 27) is reported. The greater the score, the greater the severity of depression.
Time Frame: 90 days following acute ischemic stroke
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | 20mg Dose
Number analyzed (Participants) | 32
units on a scale | 4.6 (4.1)

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | 20mg Dose
All-Cause Mortality (participants affected / at risk) | 2/34
Serious Adverse Events (participants affected / at risk) | 8/34
Other Adverse Events (participants affected / at risk) | 2/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20mg Dose (N=34)
Intermittent emesis and decreased appetite, hyponatremia serum Na+=120 mmol/L (General disorders) | 1 (1) — Intermittent emesis and decreased appetite, hyponatremia serum Na+=120 mmol/L
Abnormal lab results (General disorders) | 1 (1) — ALT=91U/L, K+=2.7mEq/L, serum Na+=139 mmol/L
Confusion, dizziness, weakness, transient aphasia (Nervous system disorders) | 1 (1) — Confusion, dizziness, weakness, transient aphasia
Right supranuclear facial palsy, left hemiparesis (Nervous system disorders) | 1 (1) — Right supranuclear facial palsy, left hemiparesis
Cardiac arrest (Cardiac disorders) | 1 (1) — Cardiac arrest
Pneumonia, severe malaria, anemia, worm infestation, and urinary tract infection (General disorders) | 1 (1) — Pneumonia, severe malaria, anemia, worm infestation, and urinary tract infection
Upper gastrointestinal bleeding, cardiac arrest (General disorders) | 1 (1) — Upper gastrointestinal bleeding, cardiac arrest
Abnormal lab results (General disorders) | 1 (1) — Hyponatremia, serum Na+=125 mmol/L
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 20mg Dose (N=34)
Urinary tract infection (Reproductive system and breast disorders) | 1 (1) — Urinary tract infection
Swelling of L arm and L foot (Skin and subcutaneous tissue disorders) | 1 (1) — Swelling of L arm and L foot

LIMITATIONS AND CAVEATS:
Our study had several limitations. There was no placebo group. Three participants were later found to lack diffuse weighted imaging (DWI) changes on brain MRI when read by an off-site neuroradiologist. We are unable to report on whether fluoxetine in combination with other interventions would be valuable or is influenced by physical therapy. Depression was not measured at enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-11-30): https://cdn.clinicaltrials.gov/large-docs/53/NCT03728153/Prot_SAP_001.pdf